CLINICAL TRIAL: NCT05006365
Title: Effects of Transcranial Pulse Stimulation (TPS) on Young Adults with Symptoms of Depression - a Pilot Randomized Controlled Trial
Brief Title: EffectsOfTranscranialPulseStimulationOnDepression-PilotRCT
Acronym: TPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HongKongPU_HSEARS20210608002
Record Dates: First submitted 2021-08-03; First posted 2021-08-16 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-09

CONDITIONS: Major Depressive Disorder
Keywords: efficacy; transcranial pulse stimulation
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcranial Pulse Stimulation (Experimental): Investigators will use a single-blind randomized controlled trial design with two-armed repeated measures. The trial design complies with the Consolidated Standards of Reporting Trials (CONSORT) statement. The first arm is the Intervention Group (Transcranial Pulse Stimulation) (TPS group)
  Interventions: Device: Transcranial Pulse Stimulation
- Waitlist Control Group (Active Comparator): Second arm is the waitlist control group.
  Interventions: Device: Transcranial Pulse Stimulation

INTERVENTIONS:
Device: Transcranial Pulse Stimulation — A total of 30 participants (both TPS group and the waitlist control group) will receive six 30 minute-TPS sessions (300 pulse in each session, total: 1800 pulse) in 2 weeks' time (i.e., 3 sessions (Monday, Wednesday, Friday) per week, total: 3 hours), on a 1: 1 allocation ratio. Participants will be followed up at 3-month period after the intervention. A 2-week TPS intervention alongside with 3-month follow-up is sufficient enough to test the effects of TPS on depressive symptoms.

SUMMARY:
The aim of this study is to evaluate the effects of transranial pulse stimulation (TPS) on young adults with symptoms of depression in Hong Kong. Methods: This is a single-blind randomized controlled trial design with two-armed repeated measures, and participants will be followed up at a 3-months post-stimulation period. Eligbility: 1) aged 18 or over; 2) able to understand/read Chinese; 3) HAM-D-17 score of ≥ 8; 4) provide written informed consent. Exclusion criteria includes: 1) individuals being prescribed a DSM-5 diagnosis other than major depressive disorder (e.g., bipolar affective disorder or schizophrenia); 2) Alcohol or substance dependence; 3) Concomitant unstable major medical conditions or major neurological conditions such as brain tumour, brain aneurysm; 4) Haemophilia or other blood clotting disorders or thrombosis; 5) Significant communicative impairments; 6) Participants with metal implant in brain or treated area of the head; 7) Participants who undertook corticosteroid treatment within the last six weeks before first TPS treatment; 8) Pregnant or breastfeeding women. Recruitment: A total of 30 subjects will be recruited from collaborative NGOs and PolyU and randomly assigned into the Intervention Group (TPS) and the Waitlist Control Group on a 1: 1 ratio. Intervention: All participants (both TPS group and the waitlist control group) will receive six 30 minute-TPS sessions (300 pulse in each session, total: 1800 pulse) in 2 weeks' time. Outcome measurements include depression, anhedonia, instrumental activities of daily living, cognition and neuroimaging.

DETAILED DESCRIPTION:
1. PRIMARY OBJECTIVE: To evaluate the effects of Transcranial Pulse Stimulation (TPS) on symptoms of depression among young adults in Hong Kong.

   SECONDARY OBJECTIVES:
2. To improve young adults' Anhedonia symptoms after the 2-week TPS intervention and will be maintained at 3-month post-intervention follow-up
3. To improve young adults' Instrumental Activities of Daily Living (IADL) after the 2-week TPS intervention and will be maintained at 3-month post-intervention follow-up.
4. To improve young adults' Cognition after the 2-week TPS intervention and will be maintained at 3-month post-intervention follow-up.
5. Post-MRI scan will show a remarkable structural and functional connectivity in participants' brain after the 2-week TPS intervention compared to pre-MRI scan.

Sample size estimation: To the best of investigator's knowledge, there is only one TPS uncontrolled pilot study conducted on 35 patients with AD in Austria and therefore, we cannot base on their effect size to estimate our sample size in this study. Considering the nature of this study is the first pilot RCT in using TPS in the treatment of depression,investigators aim at recruiting 30 subjects to evaluate the efficacy of our primary and secondary outcomes in this study.

Research plan and Methodology Methods Trial Design: In this study, the investigators will use a single-blind randomized controlled trial design with two-armed repeated measures. The trial design complies with the Consolidated Standards of Reporting Trials (CONSORT) statement. In this two-armed design, investigators will use TPS as an intervention group and a waitlist control group. A waitlist control group is appropriate for comparing the effect of the TPS on the intervention group to that of those not receiving the TPS treatment at the same timepoints Both groups will be measured at baseline (T1), immediately after the intervention (T2) and at the 3-month follow-up (T3). Based on the previous studies, a 3-month follow-up is sufficient to assess the long-term sustainability of the TPS intervention.

Intervention (Transcranial Pulse Stimulation) Purpose of the intervention: The key tenets of the TPS intervention is neuromodulation, i.e., using ultrasound-based brain stimulation techniques to modulate the human brain in a focal and targeted manner. Intervention dose: Each participant should have the pre-treatment MRI scan performed in the University Research Facility in Behavioural and Systems Neuroscience, PolyU prior coming to the first intervention session. All participants (both TPS group and the waitlist control group) will receive six 30 minute-TPS sessions (300 pulse in each session, total: 1800 pulse) in 2 weeks' time (i.e., 3 sessions (Monday, Wednesday, Friday) per week, total: 3 hours). Participants will be followed up at 3-month period after the intervention (Fig 1). The investigators believe that a 2-week TPS intervention is sufficient enough to test the effects of TPS on depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Able to understand/read Chinese
* A HAM-D-17 score of ≥ 8
* Able to provide written informed consent

Exclusion Criteria:

* Clinical Diagnosis of Major Depressive Disorder (e.g., bipolar affective disorder or schizophrenia)
* Alcohol or substance dependence
* Concomitant unstable major medical conditions or major neurological conditions such as brain tumor, brain aneurysm
* Hemophilia or other blood clotting disorders or thrombosis
* Significant communicative impairments
* Participants with metal implant in brain or treated area of the head
* Participants who undertook corticosteroid treatment within the last six weeks before first TPS treatment
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
Depression | Participants will be measured the changes of HAM-D-17 scores at baseline, immediately after intervention and at 3-months follow-up
  Hamilton Depression Rating Scale 17 (HAM-D-17) is a widely used reliable measurement. Scores range from 0 and 52, with higher scores indicating more severe depression.

SECONDARY OUTCOMES:
Anhedonia | Participants will be measured the changes of SHAPS score at baseline, immediately after intervention and at 3-months follow-up
  The core symptom of depression will be assessed by the Chinese version of the Snaith-Hamilton Pleasure Scale (SHAPS). SHAPS is a self-report scale containing 14 items. Each item scores from 1 to 4. Total scores range from 14 to 56. A higher total SHAPS score indicates lower level of anhedonia.
Instrumental Activities of Daily Living (IADL) | Participants will be measured the changes of IADL score at baseline, immediately after intervention and at 3-months follow-up
  IADL will be assessed by the 8-item Hong Kong Chinese version of the Lawton Instrumental Activities of Daily Living Scale. Each item scores from 0 or 1. Total score ranges from 0-8. A lower score indicates a higher level of dependence.
Cognition | Participants will be measured the changes of the MoCA scores at baseline, immediately after intervention and at 3-months follow-up
  Global cognition will be measured using the Hong Kong Chinese version of the Montreal Cognitive Assessment (MoCA). Montreal Cognitive Assessment is a 30-point scale, with points awarded differently depending on the type of question asked. A score between 26 to 30 indicate normal cognitive abilities. A score of 19 to 25 indicates mild cognitive impairment. Scores of between 11 and 21 suggest mild Alzheimer's disease.
Neuroimaging | Participants will be measured the changes at baseline, immediately after intervention and at 3-months follow-up
  Participants will receive pre and post treatment MRI scan to measure any changes in structural and functional connectivity changes in the brain.

CONTACTS AND LOCATIONS:
Overall Officials: Teris Cheung, PhD, Principal Investigator — HongKongPolyU
Locations (1):
- School of Nursing HongKongPolyU, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beisteiner R, Lozano AM. Transcranial Ultrasound Innovations Ready for Broad Clinical Application. Adv Sci (Weinh). 2020 Oct 27;7(23):2002026. doi: 10.1002/advs.202002026. eCollection 2020 Dec. PMID 33304757
- [Background] Hamilton M. Development of a rating scale for primary depressive illness. Br J Soc Clin Psychol. 1967 Dec;6(4):278-96. doi: 10.1111/j.2044-8260.1967.tb00530.x. No abstract available. PMID 6080235
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 Statement: Updated guidelines for reporting parallel group randomised trials. J Clin Epidemiol. 2010 Aug;63(8):834-40. doi: 10.1016/j.jclinepi.2010.02.005. Epub 2010 Mar 25. No abstract available. PMID 20346629
- [Background] Patterson B, Boyle MH, Kivlenieks M, Van Ameringen M. The use of waitlists as control conditions in anxiety disorders research. J Psychiatr Res. 2016 Dec;83:112-120. doi: 10.1016/j.jpsychires.2016.08.015. Epub 2016 Aug 21. PMID 27585425
- [Background] Liu WH, Wang LZ, Zhu YH, Li MH, Chan RC. Clinical utility of the Snaith-Hamilton-Pleasure scale in the Chinese settings. BMC Psychiatry. 2012 Oct 31;12:184. doi: 10.1186/1471-244X-12-184. PMID 23110667
- [Background] Yeung PY, Wong LLL, Chan CC, Yung CY, Leung LMJ, Tam YY, Tang LN, Li HS, Lau ML. Montreal Cognitive Assessment - Single Cutoff Achieves Screening Purpose. Neuropsychiatr Dis Treat. 2020 Nov 6;16:2681-2687. doi: 10.2147/NDT.S269243. eCollection 2020. PMID 33192067
- [Background] Graf C. The Lawton instrumental activities of daily living scale. Am J Nurs. 2008 Apr;108(4):52-62; quiz 62-3. doi: 10.1097/01.NAJ.0000314810.46029.74. PMID 18367931
- [Derived] Cheung T, Ho YS, Yeung JW, Leung SF, Fong KNK, Fong T, Kranz GS, Beisteiner R, Cheng CPW. Effects of Transcranial Pulse Stimulation (TPS) on Young Adults With Symptom of Depression: A Pilot Randomised Controlled Trial Protocol. Front Neurol. 2022 Mar 25;13:861214. doi: 10.3389/fneur.2022.861214. eCollection 2022. PMID 35401418